CLINICAL TRIAL: NCT02408068
Title: Open Label Randomised 3 Period Crossover Study to Evaluate Bioavailability of Modified Release Hydrocortisone (HC) Under Fasting & Fed Conditions & Immediate Release HC Tablets Under Fasting Conditions in Dexamethasone-suppressed Subjects
Brief Title: Effect of Slow Release Hydrocortisone on Fed & Fasting Volunteers; Immediate Release on Fasting Only
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DIUR-004
Record Dates: First submitted 2015-03-10; First posted 2015-04-03 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: subjects
MeSH Terms: interventions — Dexamethasone; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chronocort : fed (Active Comparator): Volunteers will be admitted, take dexamethasone at 22.00hrs, fast overnight, and receive a high fat, high calorie breakfast on the morning of Day 1. Thirty minutes after the start of the breakfast they will receive 20mg of modified release hydrocortisone with 200 millilitres of water, and no further food for 4 hours, water will be allowed from 1 hour after the food. Further dexamethasone doses will be given at 06:00, 12:00, 18:00 and 22:00 hours on Day 1. One baseline pharmacokinetics (PK) sample will be taken starting prior to the dose and then over 24 hours (29 samples).
  Interventions: Drug: Dexamethasone; Drug: Chronocort: fed
- Immediate release hydrocortisone: fasted (Active Comparator): Volunteers will be admitted, take dexamethasone at 22.00hrs, fast overnight, and take 20mg immediate release hydrocortisone with 200 millilitres of water on the morning of Day 1. Water will be allowed 1hr after the study drug, but no food for at least 4hrs post dose. Further dexamethasone doses will be given at 06:00, 12:00 and 18:00 hours on Day 1. One baseline pharmacokinetics (PK) sample will be taken prior to the dose, and then afterwards for over a 12 hour period (16 samples)
  Interventions: Drug: Dexamethasone; Drug: Immediate release hydrocortisone: fasted
- Chronocort: fasted (Active Comparator): Volunteers will be admitted, take dexamethasone at 22.00hrs, fast overnight, and take 20mg modified release hydrocortisone with 200millilitres of water on the morning of Day 1. Water will be allowed 1hr after the dose, but no food for at least 4hrs post dose. Further dexamethasone doses will be given at 06:00, 12:00, 18:00 and 22:00 hours on Day 1. One baseline pharmacokinetics (PK) sample will be taken prior to the dose, and then afterwards for over a 12 hour period (16 samples)
  Interventions: Drug: Dexamethasone; Drug: Chronocort: fasted

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone used to suppress endogenous cortisol secretion
Drug: Chronocort: fasted — single dose of 20mg modified release hydrocortisone in the absence of food
  Other Names: modified release hydrocortisone
  Arms: Chronocort: fasted
Drug: Immediate release hydrocortisone: fasted — single dose of 20mg immediate release hydrocortisone in the absence of food
  Other Names: Hydrocortisone
  Arms: Immediate release hydrocortisone: fasted
Drug: Chronocort: fed — single dose of 20mg modified release hydrocortisone in the presence of food
  Other Names: modified release hydrocortisone
  Arms: Chronocort : fed

SUMMARY:
The purpose of the study is to find out whether food has an effect on the way the body deals with modified release hydrocortisone, and to compare with the pharmacokinetics of immediate release hydrocortisone (fasted). This information will be used to help doctors with dosing in clinical practice.

DETAILED DESCRIPTION:
This is a phase I study in healthy male volunteers, who will be given dexamethasone to suppress their natural cortisol production. 18 will be consented for the study. They will have had a history and a physical examination, blood tests for routine safety, hepatitis C and Human Immunodeficiency Virus (HIV), drug abuse and Electrocardiograms (ECGs). Following the results of these tests and the inclusion/exclusion criteria for the study, they will be admitted to the phase I unit on the first afternoon (Day -1). They will be given dexamethasone at 22.00hrs that evening, and remain in the unit until the end of the period. Further dexamethasone doses will be given at 06:00, 12:00, and 18:00 hours on Day 1 (plus at 22:00 hours in patients given the modified release study drug). Each volunteer will be admitted for 3 periods of approximately 1.5 days, with a washout of 7 days between periods, and they will be randomised to either fast and take a single 20mg dose of immediate release hydrocortisone, to fast and take a single 20mg dose of the study medication, (a modified release hydrocortisone), or to the "fed" group, where they take a single dose of 20mg study medication, and have a highly calorific standardised breakfast. The volunteers will have cannulae to enable one pre-dose blood sample to be taken followed by 24 hour Pharmacokinetic (PK) sampling (modified release) and 12 hour PK sampling for the immediate release period. After these samples have been taken the volunteers will be able to leave the unit. There will be another assessment 3 to 5 days after study period 3 with further blood tests, assessment of any adverse events etc.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 and 60 years of age, inclusive (at screening)
* A body mass index of 21-28 (inclusive).
* No clinically significant abnormal serum biochemistry, haematology and urine examination values
* A negative urinary drugs of abuse screen. A positive alcohol test may be repeated at the discretion of the investigator.
* Negative Human Immunodeficiency Virus (HIV) and Hepatitis b & C results
* No clinically significant abnormalities in 12-lead Electrocardiogram (ECG)
* No clinically significant deviation outside the normal ranges for blood pressure and pulse measurements
* Subjects (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) and sexual partners must use effective contraception methods during the trial and for 3 months after the last dose, for example:

  * Oral contraceptive + condom
  * Intra-uterine device + condom
  * Diaphragm with spermicide + condom
* Subjects must be available to complete the study
* Subjects must provide written informed consent to participate in the study

Exclusion Criteria:

* A clinically significant history of gastrointestinal disorder likely to influence drug absorption
* Receipt of regular medication (including high dose vitamins, dietary supplements or herbal remedies)
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction Receipt of any vaccination within the previous one month
* Presence of clinically significant infections (systemic fungal and viral infections, acute bacterial infections)
* Current of previous history of tuberculosis
* A clinically significant history of previous allergy/sensitivity to hydrocortisone and/or dexamethasone
* A clinically significant history of family history of psychiatric disorders/illnesses
* A clinically significant history of drug or alcohol abuse
* Inability to communicate well with the investigator (ie language problem, poor mental development or impaired cerebral function)
* Participation in a New Chemical entity clinical study within the previous four months or a marketed drug clinical study within the previous three months
* Subjects who have consumed more than two units of alcohol pre day within seven days prior to the first dose or have consumed any alcohol within the 48hr period prior to the first dose
* Donation of greater than or equal to 450ml blood within the previous three months
* Subjects who smoke or ex-smokers who have smoked within six months prior to first dose
* Subjects who work shifts (ie regularly alternate between days, afternoons and nights)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Chronocort 20mg (fed), Chronocort 20mg (fasted), Hydrocortisone 20mg (fasted)
- Sequence 2: Chronocort 20mg (fed), Hydrocortisone 20mg (fasted), Chronocort 20mg (fasted)
- Sequence 3: Chronocort 20mg (fasted), Chronocort 20mg (fed), Hydrocortisone 20mg (fasted)
- Sequence 4: Chronocort 20mg (fasted), Hydrocortisone 20mg (fasted), Chronocort 20mg (fed)
- Sequence 5: Hydrocortisone 20mg (fasted), Chronocort 20mg (fed), Chronocort 20mg (fasted)
- Sequence 6: Hydrocortisone 20mg (fasted), Chronocort 20mg (fasted), Chronocort 20mg (fed)
Period: Treatment 1 (1.5 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment 2 (1.5 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment 3 (1.5 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross-over study so all patients received all treatments
Groups:
- All Study Participants: All patients received all 3 study treatments in randomised order
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: Chronocort Cmax
Description: Comparison of fed and fasted Chronocort Cmax for serum cortisol.
Time Frame: 24 hours
Population: PK population: All randomised subjects who had sufficient plasma concentration by time profiles for 2 adequate treatments and who did not violate the protocol in such a way that could invalidate or bias the results (major protocol violators).
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Chronocort Fed: Volunteers will be admitted, take dexamethasone to suppress endogenous cortisone at 22.00hrs and subsequently fast overnight. On the morning of Day 1, volunteers will eat a high fat breakfast and take 20mg of randomised treatment with 200 millilitres of water. Water will be allowed 1hr after the study drug is administered. One baseline pharmacokinetics (PK) sample will be taken prior to the dose, and then afterwards for over a 12 hour period (16 samples)
- Chronocort Fasted; Immediate-Release Hydrocortisone: Volunteers will be admitted, take dexamethasone to suppress endogenous cortisone at 22.00hrs, fast overnight, and take 20mg of randomised treatment with 200 millilitres of water on the morning of Day 1. Water will be allowed 1hr after the study drug, but no food for at least 4hrs post dose. One baseline pharmacokinetics (PK) sample will be taken prior to the dose, and then afterwards for over a 12 hour period (16 samples)
Arm/Group | Chronocort Fed | Chronocort Fasted | Immediate-Release Hydrocortisone
Number analyzed (Participants) | 18 | 18 | 14
nmol/L | 549.49 (17.4) | 708.46 (19.3) | 856.36 (14.6)
Statistical Analysis 1: Comparison: Chronocort Fed vs Chronocort Fasted; Results obtained using a mixed effects ANOVA with fixed effects for study period, sequence, treatment and subject (sequence) (excl. tmax); Test type: Superiority or Other; ANOVA; Geometric LSmean ratio = 77.56, 90% CI 2-sided [70.89 to 84.86]

2. Primary Outcome: Comparison of Fed and Fasted Chronocort AUC0-t
Description: Area under the curve from 0 to 24 hours for serum cortisol. Please note that the AUC0-t will be presented as a single figure (geometric mean) to represent exposure over time.
  N.B., the sampling points for Hydrocortisone are as follows: 0h, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h and 12h post-dose. However, the results for Hydrocortisone will not be incorporated into the analysis for this outcome measure.
Time Frame: 24 hours (at 0h, then 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 5.5h, 6h, 6.5h, 7h, 7.5h, 8h, 9h, 10h, 11h, 12h, 13h, 14h, 15h, 16h, 18h, 20h, 22h and 24h post-dose.)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Chronocort Fed | Chronocort Fasted | Immediate-Release Hydrocortisone
Number analyzed (Participants) | 18 | 18 | 14
h*nmol/L | 3229.26 (15.1) | 2980.85 (14.3) | 2466.90 (17.1)
Statistical Analysis 1: Comparison: Chronocort Fed vs Chronocort Fasted; Test type: Superiority or Other; ANOVA; Geometric LSmean ratio = 108.33, 90% CI 2-sided [102.30 to 114.72]

3. Primary Outcome: Comparison of Fed and Fasted Chronocort Tmax
Description: Comparison of Fed and Fasted Chronocort based on the time to achive the maximum concentration of serum cortisol
Time Frame: 24 hours
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Chronocort Fed | Chronocort Fasted | Immediate-Release Hydrocortisone
Number analyzed (Participants) | 18 | 18 | 14
hours | 6.75 (3.62) | 4.5 (1.25) | 0.87 (0.81)
Statistical Analysis 1: Comparison: Chronocort Fed vs Chronocort Fasted; Test type: Superiority or Other; p = 0.0005, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.25, 95% CI 2-sided [1.25 to 3.75]

4. Primary Outcome: Bioavailability of Chronocort® vs Hydrocortisone Tablets - Cmax
Description: Evaluation of the relative bioavailability of Chronocort® and immediate release hydrocortisone at a single dose of 20 mg in the fasted state by Cmax
Time Frame: 24 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Chronocort Fasted | Immediate-Release Hydrocortisone | Chronocort Fed
Number analyzed (Participants) | 18 | 14 | 18
nmol/L | 708.45 (19.3) | 856.36 (14.6) | 549.49 (17.4)
Statistical Analysis 1: Comparison: Chronocort Fasted vs Immediate-Release Hydrocortisone; Test type: Superiority or Other; Geometric LSmean ratio = 83.27, 90% CI 2-sided [75.58 to 91.74]

5. Primary Outcome: Bioavailability of Chronocort® vs Hydrocortisone Tablets - Fasted Using AUC0-t
Description: To evaluate the relative bioavailability of Chronocort® and immediate release hydrocortisone at a single dose of 20 mg in the fasted state using area under the curve
Time Frame: 24 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Chronocort Fasted | Immediate-Release Hydrocortisone | Chronocort Fed
Number analyzed (Participants) | 18 | 14 | 18
h*nmol/L | 2980.85 (14.3) | 2466.90 (17.1) | 3229.26 (15.1)
Statistical Analysis 1: Comparison: Chronocort Fasted vs Immediate-Release Hydrocortisone; Test type: Superiority or Other; Geometric LSmean ratio = 118.83, 90% CI 2-sided [111.58 to 126.54]

6. Primary Outcome: Bioavailability of Chronocort® vs Hydrocortisone Tablets - Fasted Using Tmax.
Description: To evaluate the relative bioavailability of Chronocort® and immediate release hydrocortisone at a single dose of 20 mg in the fasted state using Tmax.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Chronocort Fasted | Immediate-Release Hydrocortisone | Chronocort Fed
Number analyzed (Participants) | 18 | 14 | 18
hours | 4.5 (1.25) | 0.87 (0.81) | 6.75 (3.62)
Statistical Analysis 1: Comparison: Chronocort Fasted vs Immediate-Release Hydrocortisone; Test type: Superiority or Other; p = 0.0014, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 3.5, 95% CI 2-sided [2.25 to 4.38]

ADVERSE EVENTS:
Time Frame: Each study period is 1.5 days duration, so a total of 4.5 days plus a 7-day washout period between doses
Groups:
- Chronocort : Fed: Volunteers will be admitted, take dexamethasone at 22.00hrs, fast overnight, and receive a high fat, high calorie breakfast on the morning of Day 1. Thirty minutes after the start of the breakfast they will receive 20mg of modified release hydrocortisone with 200 millilitres of water, and no further food for 4 hours, water will be allowed from 1 hour after the food. One baseline pharmacokinetics (PK) sample will be taken starting prior to the dose and then over 24 hours (29 samples).
  Dexamethasone: Dexamethasone used to suppress endogenous cortisol secretion
  Chronocort: fed: single dose of 20mg modified release hydrocortisone in the presence of food
- Chronocort: Fasted: Volunteers will be admitted, take dexamethasone at 22.00hrs, fast overnight, and take 20mg modified release hydrocortisone with 200millilitres of water on the morning of Day 1. Water will be allowed 1hr after the dose, but no food for at least 4hrs post dose. One baseline pharmacokinetics (PK) sample will be taken prior to the dose, and then afterwards for over a 12 hour period (16 samples)
  Dexamethasone: Dexamethasone used to suppress endogenous cortisol secretion
  Chronocort: fasted: single dose of 20mg modified release hydrocortisone in the absence of food
- Immediate Release Hydrocortisone: Fasted: Volunteers will be admitted, take dexamethasone at 22.00hrs, fast overnight, and take 20mg immediate release hydrocortisone with 200 millilitres of water on the morning of Day 1. Water will be allowed 1hr after the study drug, but no food for at least 4hrs post dose. One baseline pharmacokinetics (PK) sample will be taken prior to the dose, and then afterwards for over a 12 hour period (16 samples)
  Dexamethasone: Dexamethasone used to suppress endogenous cortisol secretion
  Immediate release hydrocortisone: fasted: single dose of 20mg immediate release hydrocortisone in the absence of food
Arm/Group | Chronocort : Fed | Chronocort: Fasted | Immediate Release Hydrocortisone: Fasted
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 1/18 | 0/18 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronocort : Fed (N=18) | Chronocort: Fasted (N=18) | Immediate Release Hydrocortisone: Fasted (N=17)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No